CLINICAL TRIAL: NCT01685190
Title: A Randomised Phase II Trial of Prostate and pelvIs Versus prOsTate Alone Treatment for Locally Advanced Prostate Cancer
Brief Title: A Study of Prostate and pelvIs Versus prOsTate Alone Treatment for Locally Advanced Prostate Cancer
Acronym: PIVOTAL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICR-CTSU/2010/10025; CRUK/10/022 (Other Grant/Funding Number: CRUK); ISRCTN48709247 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2011-10-26; First posted 2012-09-14 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prostate Alone IMRT (Active Comparator): Participants will receive standard prostate Intensity Modulated Radiotherapy (IMRT) of 74Gy in 37 fractions delivered over 7.5 weeks.
  Interventions: Radiation: Prostate alone IMRT
- Prostate & Pelvis IMRT (Experimental): Participants will receive prostate and pelvis IMRT with a dose of 74Gy in 37 fractions delivered over 7.5 weeks to the prostate and 60Gy in 37 fractions delivered over 7.5weeks to the pelvis.
  Interventions: Radiation: Prostate and pelvis IMRT

INTERVENTIONS:
Radiation: Prostate alone IMRT — Participants will receive standard prostate IMRT of 74Gy in 37 fractions delivered over 7.5 weeks.
  Arms: Prostate Alone IMRT
Radiation: Prostate and pelvis IMRT — Participants will receive prostate and pelvis IMRT with a dose of 74Gy in 37 fractions delivered over 7.5 weeks to the prostate and 60Gy in 37 fractions delivered over 7.5weeks to the pelvis.
  Arms: Prostate & Pelvis IMRT

SUMMARY:
Prostate cancer is the most common male cancer in the UK with 35,000 cases diagnosed annually. 35% of these are locally advanced disease. These patients have a high chance of pelvic lymph node involvement and have relatively poor prostate cancer survival rates of 22.5% at 10 years.

One of the standard treatments for these patients is radiotherapy to the prostate. PIVOTAL is a multi-centre phase II non-comparative randomised feasibility trial, in which patients with a high chance of pelvic lymph node involvement are randomised between prostate radiotherapy alone and prostate + pelvic radiotherapy.

Both groups will receive radiotherapy called Intensity Modulated Radiation Therapy (IMRT). This is a relatively new method of shaping radiotherapy treatment beams which allows the tumour to be treated more precisely, whilst avoiding more of the surrounding normal, healthy tissues (particularly the rectum, bladder and bowel). Using IMRT, it is possible to deliver higher doses of radiotherapy to the pelvis than with previous radiotherapy methods - this has been tested in a single hospital, single group setting and levels of side effects (toxicity) were acceptable.

PIVOTAL aims to find out whether toxicity levels at 18 weeks from the start of radiotherapy remain acceptable when treatment is given in multiple cancer centres across the UK. It is randomised to ensure unbiased collection of acute toxicity data and to provide information on patients' willingness to participate in a randomised study. Should the phase II study be successful, the investigators would develop a phase III trial to compare treatment effectiveness (disease control).

Patients who enter PIVOTAL will be followed up for two years from the start of radiotherapy and data relating to toxicity will be collected. They will also be asked to complete patient related symptoms questionnaires. Data related to disease recurrence will then be collected annually from patients' standard hospital visits.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, non-metastatic adenocarcinoma of the prostate, previously untreated (other than by neoadjuvant hormonal treatment)
2. National Collaborative Cancer Network locally advanced disease (T3b± or T4)43 or:

   • Estimated risk of pelvic lymph node involvement ≥30% * and either:
   * Gleason 9 or 10 or
   * Gleason 8 and one other high risk feature (T3± disease or PSA >20) or
   * Gleason 7 and 2 high risk features (T3± disease and PSA ≥30)
3. WHO performance status 0 or 1
4. Normal blood count (Hb > 11g/dl, WBC >4000/mm3, platelets >100,000/mm3)
5. LHRH analogue therapy for 6-9 months duration prior to proposed radiotherapy treatment and PSA < 4ng/ml prior to randomisation.
6. Age ≥ 18 years
7. Patients must be prepared to attend follow up. All patients participating in the Patient Reported Outcomes (PRO) Study must have adequate cognitive ability to complete the PRO questionnaires.
8. Written informed consent

   * T3a disease should be demonstrated convincingly, either clinically or by MRI. T3b disease (seminal vesicle involvement) must be convincingly demonstrated on MR.

     * Risk of pelvic lymph node involvement = (Gleason score - 6) x 10 + 2/3 PSA

Exclusion criteria:

1. Prior pelvic radiotherapy
2. Prior major pelvic surgery (e.g. colectomy, colostomy, cystectomy, prostatectomy)*
3. Radiologically suspicious (short axis diameter ≥1.0cm unless biopsied and negative) or pathologically confirmed lymph node involvement
4. Life expectancy < 5 years
5. Castrate resistant prostate cancer (rising PSA after LHRHa and anti-androgen)
6. Previous active malignancy within the last 5 years other than basal cell carcinoma
7. Co-morbid conditions likely to impact on the decision to treat with radiotherapy (e.g. previous inflammatory bowel disease, previous colo-rectal surgery, significant bladder instability or urinary incontinence)
8. Bilateral hip prosthesis or fixation which would interfere with standard radiation beam configuration

   * Patients who have undergone minor pelvic surgery will be eligible (eg appendicectomy, trans urethral resection of prostate (TURP), exploratory laparoscopy, haemorrhoidectomy, inguinal/femoral hernia repair)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2011-06; Primary Completion 2013-12 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Acute lower GI RTOG toxicity at week 18 of follow-up. | 18 weeks post treatment
  Proportion of patients with acute GI RTOG grade ≥2 toxicity at week 18 from start of radiotherapy calculated as the number of patients with grade ≥2 toxicity at week 18 over the number of evaluable at week 18.

SECONDARY OUTCOMES:
Ability to deliver 60Gy in 37 fractions to the pelvis using the varying radiotherapy planning techniques and delivery systems at the participating centres. | 2 yr
Late (1 and 2 year) toxicity | 2 yr
  Measured using RTOG toxicity scale and CTCAE
Patient Reported Outcomes | 2 yr
  Participants are requested to complete questionnaires to record the impact of the treatments on bowel and bladder function.
Biochemical progression free survival | 10 yr
Time to local progression | 10 yr
Time to distant metastases | 10 yr
Overall survival | 10 yr

CONTACTS AND LOCATIONS:
Overall Officials: Prof. David Dearnaley, Principal Investigator — Institute of Cancer Research/RMHNHSFT
Locations (7):
- United Kingdom (7):
  - Queen Elizabeth, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - Velindre Hospital, Cardiff
  - Ipswich, Ipswich
  - Clatterbridge Centre for Oncology, Liverpool
  - Royal Marsden NHSFT, London
  - Freeman Hospital, Newcastle

REFERENCES:
- [Background] Harris VA, Staffurth J, Naismith O, Esmail A, Gulliford S, Khoo V, Lewis R, Littler J, McNair H, Sadoyze A, Scrase C, Sohaib A, Syndikus I, Zarkar A, Hall E, Dearnaley D; PIVOTAL Trialists. Consensus Guidelines and Contouring Atlas for Pelvic Node Delineation in Prostate and Pelvic Node Intensity Modulated Radiation Therapy. Int J Radiat Oncol Biol Phys. 2015 Jul 15;92(4):874-83. doi: 10.1016/j.ijrobp.2015.03.021. Epub 2015 Mar 30. PMID 26104940
- [Result] Dearnaley D, Griffin CL, Lewis R, Mayles P, Mayles H, Naismith OF, Harris V, Scrase CD, Staffurth J, Syndikus I, Zarkar A, Ford DR, Rimmer YL, Horan G, Khoo V, Frew J, Venkitaraman R, Hall E. Toxicity and Patient-Reported Outcomes of a Phase 2 Randomized Trial of Prostate and Pelvic Lymph Node Versus Prostate only Radiotherapy in Advanced Localised Prostate Cancer (PIVOTAL). Int J Radiat Oncol Biol Phys. 2019 Mar 1;103(3):605-617. doi: 10.1016/j.ijrobp.2018.10.003. Epub 2018 Dec 6. PMID 30528653